CLINICAL TRIAL: NCT06062225
Title: Protocol for Comparing the Efficacy of Three Reconstruction Methods of the Digestive Tract (Kamikawa Versus Single-Tract Jejunal Interposition Versus SOFY Reconstruction) After Proximal Gastrectomy
Brief Title: Protocol for Comparing the Efficacy of Three Reconstruction Methods of the Digestive Tract After Proximal Gastrectomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Changzhi People's Hospital Affiliated to Changzhi Medical College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020TD27
Record Dates: First submitted 2023-09-25; First posted 2023-10-02 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-09

CONDITIONS: Proximal Gastric Adenocarcinoma; Gastrectomy; Anastomosis; Reflux Esophagitis; Postoperative Complications
MeSH Terms: conditions — Esophagitis, Peptic; Postoperative Complications

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Kamikawa reconstruction (Experimental): Patients will be administered Kamikawa reconstruction after proximal gastrectomy.
  Interventions: Procedure: Kamikawa
- STJI reconstruction (Active Comparator): Patients will be administered Single-Tract Jejunal Interposition(STJI) reconstruction after proximal gastrectomy.
  Interventions: Procedure: STJI
- SOFY reconstruction (Active Comparator): Patients will be administered SOFY reconstruction after proximal gastrectomy.
  Interventions: Procedure: SOFY

INTERVENTIONS:
Procedure: Kamikawa — Kamikawa reconstruction after proximal gastrectomy
  Arms: Kamikawa reconstruction
Procedure: STJI — Single-Tract Jejunal Interposition(STJI) reconstruction after proximal gastrectomy
  Arms: STJI reconstruction
Procedure: SOFY — SOFY reconstruction after proximal gastrectomy
  Arms: SOFY reconstruction

SUMMARY:
The efficacy of three different reconstruction methods after proximal gastrectomy will be investigated in this study through a prospective, multicenter, randomized controlled trial.

DETAILED DESCRIPTION:
In the trial, 180 patients with proximal early gastric cancer will be enrolled and then randomly assigned to one of three groups: Group A (Kamikawa, n = 60), Group B (single-tract jejunal interposition, n = 60), or Group C (SOFY reconstruction, n = 60). The general information, past medical history, laboratory and imaging findings, and surgical procedures of each patient will be recorded. Patients in Group A, Group B and Group C will receive Kamikaze reconstruction, single-tract jejunal interposition reconstruction and SOFY reconstruction respectively after standard proximal gastrectomy and lymph nodes dissection. The primary endpoint will be the incidence of reflux esophagitis, while the incidence of anastomotic leakage, anastomotic stenosis, operative time, and intraoperative blood loss will be secondary endpoints to compare the efficacy of these three reconstruction methods after proximal gastrectomy.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20-75 years old, male or female;
* Pathological diagnosis of preoperative endoscopic biopsy: the tumor is located in the upper 1/3 of the stomach (including the esophagogastric junction), and the clinical staging of gastric cancer： Ia and Ib (T1N0M0, T1N1M0, and T2N0M0) (14) according to the eighth edition of the AJCC (15);
* No distant metastasis observed on preoperative chest radiograph, abdominal ultrasound or upper abdominal CT;
* ASA grade 1-3;
* Patients without contraindications to surgery;
* Patients and their families voluntarily signing the informed consent form and participating in the study;

Exclusion Criteria:

* Patients diagnosed with primary tumors or distant metastasis;
* Patients whose tumor is located in the greater curvature side of the stomach;
* Patients with coagulation dysfunction which could not be corrected;
* Patients who were diagnosed with viral hepatitis and cirrhosis;
* Patients who were diagnosed with diabetes mellitus, uncontrolled or controlled with insulin;
* Patients with organ failure such as heart, lung, liver, brain, kidney failure;
* Patients with ascites or cachexia preoperatively in poor general conditions;
* Patients diagnosed with immunodeficiency, immunosuppression or autoimmune diseases (such as allogeneic bone marrow transplant, immunosuppressive drugs, SLE, etc.).
* Patients refusing to sign the informed consent of the study;

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
incidence of reflux esophagitis | 24 months after surgery
  The percentage (%) of patients developing postoperative reflux esophagitis after surgery in each group.

SECONDARY OUTCOMES:
incidence of anastomotic leakage | 14 days after surgery
  The percentage (%) of patients developing postoperative anastomotic leakage after surgery in each group.
incidence of anastomotic stenosis | 24 months after surgery
  The percentage (%) of patients developing anastomotic stenosis after surgery in each group.
operative time | 1 day after surgery
  The duration, measured in minutes, spent on reconstructing the digestive tract using specific method (Kamikawa, STJI or SOFY) following proximal gastrectomy.
intraoperative blood loss | 1 day after surgery
  The amount of blood, measured in milliliters, lost during the reconstruction of digestive tract using specific method (Kamikawa, STJI or SOFY) following proximal gastrectomy.

CONTACTS AND LOCATIONS:
Overall Officials: Wenqing Hu, Study Chair — Changzhi People's Hospital Affiliated to Changzhi Medical College

IPD SHARING:
Plan to Share IPD: No